CLINICAL TRIAL: NCT06475352
Title: Dihydropyrimidine Dehydrogenase (DPD) Phenotype-guided Dose Individualization of Fluoropyrimidine-based Chemotherapy in DPD Deficient Patients With Gastrointestinal Cancers
Brief Title: Dose Individualization of Chemotherapy in Patients With Gastrointestinal Cancers Lacking a Specific Liver Enzyme
Acronym: FUDOSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-2311; 2023-509963-25-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Digestive Cancer; Colorectal Cancer
Keywords: Fluoropyrimidine; FOLFOX; CAPOX; Adjuvant; Metastatic; Recurrent; Colorectal; digestive; Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis; Recurrence; Neoplasms | interventions — Folfox protocol; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Uracilemia <16 (Active Comparator): Patient with uracilemia <16 ng/mL will receive a full standard fluoropyrimidine dose
  Interventions: Drug: FOLFOX regimen; Drug: CAPOX regimen
- Uracilemia [16-20[ (Experimental): Patients with uracilemia between [16-20[ ng/mL will receive a full standard fluoropyrimidine dose -dose
  Interventions: Drug: FOLFOX regimen; Drug: CAPOX regimen
- Uracilemia [20-50[ - 25% (Experimental): Patients with uracilemia between [20-50[ ng/mL will be randomized to receive a 25% fluoropyrimidine dose reduction
  Interventions: Drug: FOLFOX regimen; Drug: CAPOX regimen
- Uracilemia [20-50[ - 50% (Experimental): Patients with uracilemia between [20-50[ ng/mL will be randomized to receive a 50% fluoropyrimidine dose reduction
  Interventions: Drug: FOLFOX regimen; Drug: CAPOX regimen
- Uracilemia [50-100[ (Experimental): Patients with uracilemia between [50-100[ ng/mL will receive a 50% fluoropyrimidine dose reduction
  Interventions: Drug: FOLFOX regimen; Drug: CAPOX regimen
- Uracilemia [100-150[ (Experimental): Patients with uracilemia between [100-150[ ng/mL will receive a 75% fluoropyrimidine dose reduction
  Interventions: Drug: FOLFOX regimen; Drug: CAPOX regimen

INTERVENTIONS:
Drug: FOLFOX regimen — Oxaliplatin will be administered at a fixed dose of 85 mg/m² by 2h intravenous (IV) infusion concurrently with folinic acid 400 mg/m² (or 200 mg/m² if L-folinic acid) as a 2 h IV infusion on day 1 of each 14-day cycle followed by 5-fluorouracil (5-FU) 400 mg/m² IV bolus on day 1, then continuous IV infusion of 1,200 mg/m² /day × 2 days (total 2400 mg/m² for 46-48 hours)
Drug: CAPOX regimen — Oxaliplatin will be administered at a fixed dose of 130 mg/m² by 2h IV infusion on day 1 of each 21-day cycle followed by capecitabine (1000 mg/m²) twice a day (BID) during 2 weeks, every 3 weeks

SUMMARY:
The goal of this clinical trial is to establish guidelines for fluoropyrimidine dose reduction according to uracilemia in patients with DPD deficiency in the treatment of digestive cancers. The main question it aims to answer is:

- Which reduction dose of fluoropyrimidine is needed for patient with DPD deficiency?

Participants will:

* Take the treatment with the reduction of dose stated by the protocol
* Visit the clinic once every 2-3 weeks for checkups and tests for collection of adverse events

DETAILED DESCRIPTION:
Multicenter phase II trial evaluating different strategies of pre-specified fluoropyrimidine-dose adjustment according to [U] in DPD-deficient patients with gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pre-treatment screening based on [U] value according to INCa/HAS recommendations.
2. Eastern Cooperative Oncology Group performance status (ECOG PS) ≤2
3. Fluoropyrimidine-naïve patients with gastrointestinal cancer starting chemotherapy combining fluoropyrimidine (5-FU or capecitabine) and oxaliplatin whatever the context (adjuvant, neoadjuvant, palliative) including the following regimens (the most frequently prescribed in gastrointestinal cancers):

   * biweekly 5-FU and oxaliplatin (FOLFOX) +/- targeted therapy (TT)
   * three-weekly capecitabine and oxaliplatin (CAPOX) +/- TT
4. Age ≥ 18 years
5. Patients eligible for full standard fluoropyrimidine and oxaliplatin doses regardless of DPD deficiency
6. Adequate bone marrow function (cell blood count (CBC)), estimated glomerular filtration rate (DFG) ≥ 50 ml/min, alkaline phosphatase (ALP) / aspartate aminotransferase (ASAT) / alanine aminotransferase (ALAT) ≤ 5 upper limit of normal (ULN), and bilirubin ≤ 50 micromol/L
7. Patient must have signed and dated a written informed consent form prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
8. Women of childbearing potential must have a negative serum or urine pregnancy test.
9. Patients must agree to remain abstinent or use contraceptive methods with a failure rate of < 1% per year for the duration of study treatment and within 6 months after completing treatment.
10. Patients must be affiliated to a Social Security System (or equivalent).
11. Patient is willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.

Exclusion Criteria:

1. Patients with complete DPD deficiency based on [U] ≥150 ng/mL
2. Any prior treatment including a fluoropyrimidine
3. Patients with any contraindication to treatment with fluoropyrimidine or oxaliplatin regardless of DPD deficiency
4. Patients not eligible for full standard dose fluoropyrimidine and oxaliplatin for clinical reasons including older age and/or comorbidity regardless of a DPD deficiency
5. Patients unwilling or unable to comply with trial obligations for geographic, social, or physical reasons, or who are unable to understand the purpose and procedures of the trial
6. Recent or concomitant treatment with brivudine
7. Pregnant or breastfeeding woman.
8. Participation in another therapeutic trial within 30 days prior to inclusion.
9. Persons deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of fluoropyrimidine-induced grade ≥ 3 haematological and gastrointestinal toxicity after 2 cycles | Throughout the two first cycles of treatment, up to 42 days
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.

SECONDARY OUTCOMES:
Recommended fluoropyrimidine dose | Throughout the four first cycles of treatment, up to 3 months
  The rate of fluoropyrimidine induced grade ≥ 3 haematological and gastrointestinal toxicity in each uracilemia-based group of DPD-deficient patients (according to uracilemia level) compared to the rate observed in non DPD-deficient patients (control arm)
Description of fluoropyrimidine dose | Throughout the four first cycles of treatment, up to 3 months
  The cumulative dose (mg/m²) of chemotherapy delivered to patients will be recorded along with reasons of dose-modifications or treatment discontinuation for limiting toxicity
Percentage of fluoropyrimidine dose modification | Throughout the four first cycles of treatment, up to 3 months
  Percentage of patients for whom fluoropyrimidine dose is increased or decreased
Fluoropyrimidine toxicity during the study | Throughout the four first cycles of treatment, up to 3 months
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Disease-free survival (DFS) - Stage III Colon Cancer | 3 years
  Disease-free survival is defined as the delay between date of inclusion and tumor relapse (local, regional, or distant) or death from any cause, whichever occurs first.
Overall survival (OS) - Stage III Colon Cancer | From randomization to death from any cause, up to 3 years.
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Progression-free survival (PFS) - Stage IV Colon Cancer | From randomization to disease progression or death, up to 1 year.
  The progression-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BOIGE, MD, Principal Investigator — Gustave Roussy Cancer Campus; Marie-Anne LORIOT, Study Director — Hopital Europeen Georges Pompidou
Locations (34):
- France (34):
  - CHU Amiens, Amiens
  - Institut du Cancer Avignon Provence, Avignon
  - CH Aunay Bayeux, Bayeux
  - CH Cote Basque, Bayonne
  - CHU Besançon, Besançon
  - Centre François Baclesse, Caen
  - Polyclinique du Parc - Centre d'Oncologie Maurice Tubiana, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Hopital Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - GH Mutualiste de Grenoble, Grenoble
  - Hopital Privé Drome-Ardeche, Guilherand-Granges
  - CHU Dupuytren, Limoges
  - Hopital Privé Jean Mermoz, Lyon
  - Centre Léon Bérard, Lyon
  - Grand Hopital de l'Est Francilien, Meaux
  - Hopital Nord Franche Comté - Site du Mittan, Montbéliard
  - Centre Antoine Lacassagne, Nice
  - CHU d'Orléans, Orléans
  - Institut Curie, Paris
  - Hopital Saint Louis, Paris
  - Hopital Saint Antoine, Paris
  - GH Diaconesses Croix St Simon, Paris
  - CHU Bordeaux, Pessac
  - Hospices Civiles de Lyon, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Hopital Robert Debré, Reims
  - Institut Jean Godinot, Reims
  - CH de Saint Malo, St-Malo
  - Institut du Cancer de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - Hopital Bretonneau, Tours
  - Gustave Roussy Cancer Campus, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.